CLINICAL TRIAL: NCT02193503
Title: An Open Phase I Clinical Study Assessing Safety and Tolerability of MVX-ONCO-1 in Patients With Solid Tumor Who Are Not/Not Any Longer Amenable to Standard Therapy
Brief Title: MVX-ONCO-1 in Patients With Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Maxivax SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVX-2011-01
Record Dates: First submitted 2013-08-26; First posted 2014-07-17 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor; Cancer
Keywords: cancer; solid tumors; gene therapy; cell therapy; encapsulation
MeSH Terms: conditions — Neoplasms | interventions — Therapeutics; Equipment and Supplies; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): MVX-1-loaded capsules and injection of irradiated autologous tumor cells
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Treatment is the implantation of loaded capsules + injection of irradiated autologous tumor cells
  Other Names: - capsules MVX-1-loaded (medical device); - irradiated autologous tumor cells (cell therapy)

SUMMARY:
The objectives are to assess the safety and tolerability of 6 vaccine doses of MVX-ONCO-1, administered sub-cutaneously (injections and capsules implantations), in patients with advanced metastatic solid tumor in progression who are not or not any longer amenable to any standard therapy of their tumour disease.

DETAILED DESCRIPTION:
Endpoints:

Primary: To assess safety parameters including adverse and serious adverse events (incidence, causality, severity), local and systemic tolerance to the administered study treatment, changes in laboratory values and vital signs in patients with solid tumor; Secondary: to measure some tumor responses in using imaging technique, serological tumor markers, immune monitoring and metabolic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years and older with advanced metastatic cancer in progression of various sites [Carcinoma of lung (either small cell or non-small cell), colon, breast, pancreas (exocrine or endocrine), stomach, oesophagus, head&neck, thyroid, kidney, bladder, prostate, ovary, uterus (cervix or corpus); Sarcoma of soft tissue, bone, uterus, melanoma; primary brain tumor] where all recognized treatment are exhausted or not feasible.
* Life expectancy: estimate of at least 4 months.

Exclusion Criteria:

* Have participated in any other investigational study or received an experimental therapeutic procedure considered to interfere with the study in the 4 preceding weeks.
* Have received any chemotherapy treatment in the 4 preceding weeks.
* Serious concomitant health condition such as organ transplant requiring immunosuppressive drugs, severe psychiatric disorders.
* History of second cancer within the last 2 years with the exception of basal cell carcinoma of skin and localized cervical carcinoma treated with curative intent.
* Patient with a systemic disease other than cancer, that is not controlled by usual medication.
* Therapeutic anticoagulation with coumarine or continues iv heparin. Low-molecular weight heparin (LMWH) is permitted as long as treatment can be withheld several hours prior to subcutaneous implantation.
* Positive HIV-1, HIV-2, HTLV-1, HTLV-2, hepatitis B surface antigen, or hepatitis C antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events and/or Serious Adverse Events | 18 weeks
  Adverse events will be followed carefully at each clinic visit by the Investigator, to determine their incidence, causality and severity.

SECONDARY OUTCOMES:
Delayed type hypersensitivity reactions, Induction of a specific CD8 response | 18 weeks
  immune monitoring
imaging and metabolic monitoring | 18 weeks
tumor size | 18 weeks
  document of tumor number, sites, size of lesions
tumor pain | 18 weeks
  intensity, site, frequency of pain, use of analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Fernandez, MD, Principal Investigator — HUG
Locations (1):
- Hopitaux Universitaires de Genève - HUG, Geneva, Canton of Geneva, Switzerland